CLINICAL TRIAL: NCT01337115
Title: Effect of a Single Shot Sciatic Nerve Block (SNB) Combined With a Continuous Femoral Block (CFNB) on Pain Scores After Knee Arthroplasty. A Randomized Controlled Trial
Brief Title: Effect of a Sciatic Block (SNB) Combined With a Continuous Femoral Block (CFNB) on Pain Scores After Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Raul Carvalho, Anesthesiology Consultant, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA 007/11(004-DEFI/007-CES)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Knee arthroplasty; Peripheral nerve blocks; Sciatic nerve block; Femoral nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous femoral nerve block (CFNB) (Active Comparator): A continuous femoral nerve block is performed for peri-operative analgesia and a bolus of 30 ml of ropivacaine 0.375% is injected before induction of general anesthesia and surgery starts. An infusion of 8ml/h of ropivacaine 0.2% is started in post anesthesia care unit (PACU) and maintained for 48h
  Interventions: Procedure: CFNB
- Single shot SNB plus CFNB (Experimental): A single shot sciatic nerve block (SNB) is performed before surgery with 25ml of 0.2% ropivacaine in addition to the continuous femoral nerve block (CFNB) performed in the control group before induction of general anesthesia and surgery starts. An infusion of 8ml/h of ropivacaine 0.2% is started in Post anesthesia care unit (PACU) and maintained for 48h
  Interventions: Procedure: SNB plus CFNB

INTERVENTIONS:
Procedure: SNB plus CFNB — A single shot sciatic nerve block (SNB) is performed with 25 ml of 0.2% ropivacaine before surgery in addition to an isolated continuous femoral nerve block (CFNB) in the control group
  Other Names: Peripheral nerve blocks; Local anesthetics; Ropivacaine; Femoral nerve block; Sciatic nerve block
  Arms: Single shot SNB plus CFNB
Procedure: CFNB — A continuous femoral nerve block is performed for peri-operative analgesia and a bolus of 30 ml of ropivacaine 0.375% is injected before induction of general anesthesia and surgery starts. An infusion of 8ml/h of ropivacaine 0.2% is started in post anesthesia care unit (PACU) and maintained for 48h
  Other Names: Peripheral nerve blocks; Local anesthetics; Ropivacaine; Femoral nerve block
  Arms: Continuous femoral nerve block (CFNB)

SUMMARY:
The purpose of this study is to determine if the addition of a sciatic nerve block (SNB) to a continuous femoral nerve block (CFNB) improves post-operative analgesia after knee arthroplasty.

DETAILED DESCRIPTION:
Background: Postoperative pain after total knee replacement /arthroplasty (TKA) is a major concern. It is severe pain in 60% of patients and moderate in 30%. Continuous femoral nerve blocks (CFNB) are considered an excellent choice for regional anesthesia for major knee repair but there are some controversies about the need of supplemental obturator or sciatic nerve blocks for achieving better postoperative analgesia. A recent meta-analysis states there is no sufficient evidence to recommend or discharge these associations.

Objectives: We aim to assess the efficacy of the association of a sciatic nerve block (SNB) and a continuous femoral nerve block (CFNB) for reducing postoperative pain in patients submitted to TKA. Methods: A randomized controlled study on 50 patients submitted to TKA. Control group receives a femoral nerve block with a catheter before general anesthesia is induced and the intervention group gets a similar block plus a single shot SNB before general anesthesia. Both groups start a continuous local anesthetic infusion through femoral catheter after the end of surgery and supplemental oral diclofenac and paracetamol. Pain scores are measured until 24h postoperatively, side effects and patient satisfaction are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral total knee replacement

Exclusion Criteria:

* Contra-indication for general anesthesia
* Infection on puncture site
* Coagulation disorders
* Pre-existent neuropathies
* Allergies to local anesthetics, paracetamol, diclofenac and tramadol
* Severe dyspepsia
* Less than 50kg weigh
* Body Mass Index (BMI) greater than 40
* American Society of Anesthesiologists (ASA) Physical Status 4 or 5
* Absence of capacity to use the Visual Analog Score (VAS) scale
* Refusal to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul MS Carvalho, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Serviço de Anestesia, Porto, Porto District, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2011-February 2012. Consecutive patients for total knee arthroplasty at Orthopedic Department, Centro Hospitalar do Porto
Pre-assignment Details: Patients were excluded before randomization if refuse, could not use Visual Analogue Scale (VAS) scale, had contraindications for any of the components of the anesthesia protocol or, anesthesiologist was not expert in peripheral blocks
Groups:
- Continuous Femoral Nerve Block (CFNB): A continuous femoral nerve block is performed for peri-operative analgesia and a bolus of 30 ml of ropivacaine 0.375% is injected before surgery starts. An infusion of 8ml/h of ropivacaine 0.2% is started in PACU and maintained for 48h
- Single Shot Sciatic Nerve Block (SNB): A single shot sciatic nerve block is performed before surgery with 25ml of 0.2% ropivacaine in addition to the continuous femoral nerve block performed in the control group
Period: Overall Study
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB)
Started | 25 | 25
Completed | 23 (2 patients could not be assessed after 12h because of catheter dislocation) | 25
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 25
  >=65 years | 15 | 10 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 68.16 (9.83) | 65.44 (8.93) | 66.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  Portugal | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scores (VAS) - Pain Scores Measured in mm (0-100)
Description: Pain scores measured by Visual Analogue Score (VAS) scale at 15-30min after Post anesthesia care unit (PACU) arrival VAS is a 100mm scale to measure pain. 0mm - no pain 100mm - worst possible pain
Time Frame: 15-30 min after arrival on post anesthesia care unit (PACU)
Population: Participants were analyzed in an Intention to treat (ITT) manner. All randomized subjects (25 in each arm) completed the protocol so all were included for analysis as planned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB)
Number analyzed (Participants) | 25 | 25
units on a scale | 59.4 (27.2) | 30.2 (30.5)
Statistical Analysis 1: Comparison: Continuous Femoral Nerve Block (CFNB) vs Single Shot Sciatic Nerve Block (SNB); Difference between mean VAS pain scores. Power 80%. Null hypothesis states there is no difference between pains scores in both groups; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 28.44, 95% CI 2-sided [11.55 to 45.34], Standard Error of Mean 8.4

2. Secondary Outcome: Satisfaction With Anesthesia Technique in Each Arm of the Study
Description: Satisfaction with the anesthesia technique using a categorical scale with three levels:
  Bad Reasonable Good/Very Good A Fisher's Exact test is made to asses any differences in the distribution of patients in each arm to each level of the categorical scale
Time Frame: 1 month after surgery
Population: Analysis was performed on Participants available for telephone contact one month after surgery and was made per protocol.
Measure: Number; unit: participants
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB)
Number analyzed (Participants) | 20 | 21
participants
  Bad | 0 | 0
  Reasonable | 3 | 2
  Good/Very Good | 17 | 11
Statistical Analysis 1: Comparison: Continuous Femoral Nerve Block (CFNB) vs Single Shot Sciatic Nerve Block (SNB); Test type: Superiority or Other; p = 0.537, Fisher's exact test — The null hypothesis is that there is no difference in patient satisfaction distribution by the three categories used (Bad; Reasonable; Good/Very Good) between groups; Fisher's Exact test allows to test for the significance of the distribution in the results table with three categories

3. Primary Outcome: VAS Results - Pain Measured in mm (0-100)
Description: VAS pain scores are measured by blinded investigators 12h after surgery .
  VAS scale:
  0 - no pain 100 - worst possible pain
Time Frame: 12h after surgery
Population: All 25 patients in each arm completed the protocol. Analysis was made in an ITT manner.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CFNB: Patients with continuous femoral nerve block
- CFNB+Single Shot SNB: Patients with additional sciatic nerve block
Arm/Group | CFNB | CFNB+Single Shot SNB
Number analyzed (Participants) | 25 | 25
units on a scale | 26.1 (23.8) | 9.2 (14.8)
Statistical Analysis 1: Comparison: CFNB vs CFNB+Single Shot SNB; Null hypothesis states that there is no difference between groups. Power 80%; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Median Difference (Final Values) = 16.92, 95% CI 2-sided [5.52 to 28.33], Standard Error of Mean 5.67

4. Primary Outcome: VAS Results - Pain Scores Measured in mm (0-100)
Description: VAS pain scores are measured by blinded investigators 24h after surgery .
  VAS scale:
  0 - no pain 100 - worst possible pain
Time Frame: 24h after surgery
Population: In the CFNB group 2 patients did not complete the protocol. Analysis was made in an ITT manner and Last Observational Carried Forward (LOCF) was the imputation technique used. In the SNB group, all 25 patients completed the protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB)
Number analyzed (Participants) | 23 | 25
units on a scale | 30.13 (24.97) | 32.68 (24.49)
Statistical Analysis 1: Comparison: Continuous Femoral Nerve Block (CFNB) vs Single Shot Sciatic Nerve Block (SNB); Null hypothesis states there is no difference between both groups. Power 80% to detect 15% difference in means; Test type: Superiority or Other; p = 0.723, t-test, 2 sided; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-16.93 to 11.83], Standard Error of Mean 7.14

ADVERSE EVENTS:
Time Frame: 24h
Description: Motor block, paresthesias, falls or serious nausea and vomiting were monitored
Arm/Group | Continuous Femoral Nerve Block (CFNB) | Single Shot Sciatic Nerve Block (SNB)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Difficulties in contacting patients by phone and getting reliable answers limit the value of the patient satisfaction parameter.

No analysis was made on the effect of nerve blocks on rehabilitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes